CLINICAL TRIAL: NCT00418197
Title: A Prospective and Randomized Controlled Trial to Evaluate the Safety and Effectiveness of Total Facet Arthroplasty in the Treatment of Degenerative Spinal Stenosis
Brief Title: Total Facet Arthroplasty System®(TFAS®) Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Archus Orthopedics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR0051
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Spinal Stenosis; Low Back Pain; Spondylolisthesis; Lumbar Spinal Stenosis; Leg Pain; Spinal Diseases
Keywords: spinal stenosis; low back pain; spondylolisthesis; lumbar spinal stenosis; leg pain; spinal diseases
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain; Spondylolisthesis; Spinal Diseases

INTERVENTIONS:
Device: Total Facet Arthroplasty System® (TFAS®)

SUMMARY:
The Archus Total Facet Arthroplasty System® (TFAS®) is a non-fusion spinal implant indicated for treatment of patients with moderate to severe spinal stenosis. TFAS® replaces the diseased facets following surgical removal. TFAS® offers the surgeon new options for treating spinal stenosis patients, enabling a more comprehensive decompression via complete removal of the facets. TFAS® also offers an alternative to rigid spinal fusion fixation enabling intervertebral motion. The clinical trial is intended to demonstrate restoration of stability and sagittal balance to the spine. TFAS® also eliminates the need for painful bone graft harvest from the patient's hip which may be required with fusion procedures.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative spinal stenosis, central or lateral, at spinal levels L3-L4 or L4-L5
* Skeletally mature male or female between the ages of 50 and 85 years of age inclusive
* No greater than Grade I degenerative spondylolisthesis at the index level
* Persistent leg symptoms,including pain, numbness, burning or tingling for a minimum duration of six months
* Operative candidates with no more than three levels of degenerative lumbar spinal stenosis requiring decompression
* Failed to respond to non-operative treatment modalities for a minimum duration of six months

Exclusion Criteria:

* Male or female less than 50 or greater than 85 years old Grade 2 or higher spondylolisthesis or any retrolisthesis at the index level
* More than 3 vertebral levels of degenerative spinal stenosis requiring decompression
* More than 1 vertebral level of degenerative spinal stenosis requiring instrumentation
* Not available for long term follow-up and interval visits
* Prior or concurrently planned lumbar fusion or disc replacement at any level of the lumbar spine
* Two or more previous surgeries to the lumbar spine at the same level to be implanted
* Is being treated with other devices for the same disorder (e.g. pain control devices)
* Active systemic infection or infection at the operating site
* Osteoporosis
* Known sensitivity to device materials
* Has an immunosuppressive disorder
* Has a medical condition that may interfere with clinical evaluations
* Is obese defined by a patient body mass index greater than 40
* Has significant scoliosis (Cobb >25°)
* Is pregnant or planning to become pregnant within the proposed three year investigation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2005-08

PRIMARY OUTCOMES:
The primary safety and efficacy evaluation endpoints to determine individual patient success are the Zurich Claudication Questionnaire (ZCQ), neurologic status, solid fusion for the control (spinal fusion) group.

SECONDARY OUTCOMES:
Visual Analog Scales (VAS) for Leg and Back pain, SF-36 scores, radiographic measurements.